CLINICAL TRIAL: NCT03536468
Title: Short Term Psychological Impact of Tooth Loss in Patients Consulting in a University Dental Clinic
Brief Title: Psychological Impact of Tooth Loss
Acronym: Edentpsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17037J
Record Dates: First submitted 2018-04-13; First posted 2018-05-24 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2018-11

CONDITIONS: Edentulous Mouth; Partial Edentulism
Keywords: Tooth loss, edentulousness, psychology, oral health-related
MeSH Terms: conditions — Mouth, Edentulous; Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients pending complete tooth loss: Will be recruited patients pending tooth loss, ages between 18 and 65 years, whose dental conditions have previously been identified

SUMMARY:
Tooth loss impact on daily living, mood and self-perceived well-being. However, psychological impact of teeth loss has not been evaluated. Present study aims to evaluate the psychological conditions of patients pending complete tooth extraction before and shortly after tooth loss using Hospital Anxiety and Depression scale (HAD) and Geriatric Oral Health Assessment Index (GOHAI).

DETAILED DESCRIPTION:
Patients will be interviewed concerning their psychological conditions (HADS) and their oral health related quality of life (GOHAI) before tooth extraction and one month after complete tooth loss.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate to the study
* dental status identified

Exclusion Criteria:

* uncooperative ou patient not able to complete the questionary
* adult patients under protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients pending complete tooth extraction within the groupe hospitalier Pitie Salpétrière
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital anxiety and depression (HAD) score | 1 month (change in score from baseline (before tooth extraction) to 1 month after tooth extraction)
  The HADS is a 14-item self-assessment scale designed to evaluate emotional stress induced by chronic pain in non-psychiatric populations. HAD-A assessed anxiety and HAD-D evaluated depression. Scores of greater than 10 were indicative of anxiety or depression, scores of 7 or less were indicative of no significant anxiety and depression, and scores of 8 to 10 indicated borderline anxiety or depression.

SECONDARY OUTCOMES:
Change in General oral health assessment index (GOHAI) | 1 month (change in score from baseline (before tooth extraction) to 1 month after tooth extraction)
  The General oral health assessment index (GOHAI) is a questionnaire about the impact of oral health on quality of life. It includes 12 items evaluating three dimensions of oral health with respect to quality of life: (1) functional field (eating, speaking, and swallowing); (2) psychological field (appearance, social relationship); (3) pain or discomfort concerning gums or teeth. Each item has a score ranging from 1 to 5. The GOHAI-add score corresponds to the sum of the scores and ranges from 12 to 60 (20 for functional field, 25 for psychological field, and 15 for comfort/pain field). A score higher than 57 is high and indicates a satisfactory oral quality of life. A score from 51 to 56 is average and a score of 50 or less is low, reflecting a poor oral quality of life.
Gender | at date of inclusion (up to 24h)
  Respondents complete a questionnaire identifying their gender (man or woman)
Age | at date of inclusion (Up to 24h)
  Respondents complete a questionnaire identifying their age (in years)
Educational level | at date of inclusion (Up to 24h)
  Respondents complete a questionnaire identifying their educational level : last degree (no degree at al, French General Certificate Secondary Education, High School Diploma, Vocational Training Certificate taken at Secondary School, university degree)
Income | at date of inclusion (Up to 24h)
  Respondents completed a questionnaire identifying their income level each month (in euros)
General health | at date of inclusion (Up to 24h)
  Respondents complete a questionnaire indentifying their general heath and the existence of disease
Dental status | at date of inclusion (Up to 24h)
  Dental Examination is done by a dental practioner

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Braud, Study Director — APHP
Locations (1):
- Pôle odontologie Hôpital Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided